CLINICAL TRIAL: NCT04480177
Title: Effect of Intrinsic Foot Muscles Training and Foot Orthosis on the Medial Longitudinal Arch in Flexible Flatfoot Subjects
Brief Title: Effect of Foot Muscles Training and Foot Orthosis on the Medial Arch in Flatfoot Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shaikha Uthman, master student, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGS-2018-03-184
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Flexible Flatfoot
Keywords: Flatfoot; Insole; Short-foot exercise; Orthotic
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insole group (Other): the control group receives insole only.
  Interventions: Device: foot insole
- exercise group (Experimental): the experimental group receives exercise and insole.
  Interventions: Device: foot insole; Other: short foot exercise

INTERVENTIONS:
Device: foot insole — the subject was instructed to wear foot insole for 8 hours.
Other: short foot exercise — the subject was instructed to perform exercise once a day 30 repetitions.
  Arms: exercise group

SUMMARY:
Orthotic therapy or exercise therapy is the standard conservative treatment for flexible flat foot. Little is known about the effectiveness of their interaction on managing flatfoot.

The study aims to evaluate the effect of insoles and short foot exercise on the height and area of the medial longitudinal arch of flexible flatfoot participants as well as the force and pressure.

DETAILED DESCRIPTION:
Study design: A parallel, active-control study design was used to conduct a single-blinded randomized controlled trial.

Method: The toe rising test, the "too many toes" sign, and the navicular drop test was used to select 30 participants with flexible flatfoot. Participants was randomly assigned either to an experimental group (n = 15) or a control group (n = 15). The experimental group received short foot exercises (SFE) and insoles, and the control group received only insoles. SFE was implemented 30 times for a duration of three minutes each day over the course of six weeks. The exercise progressed from sitting to standing and finally to one leg stance position within every two weeks. The participants wore shoes containing orthotic insoles for eight hours per day for six weeks. The EMED-x system was used to measure plantar pressure distribution (force, area, and pressure) at baseline and at two-week intervals throughout the six-week intervention. The Lower Extremity Functional Scale (LEFS) was used to evaluate restriction in participants' functional abilities, and the navicular drop test (NDT) was used to assess the medial longitudinal arch (MLA) height. Both variables were measured at baseline and at the sixth week.

Statistics: Mixed-effects ANOVA was used to test for significant interactions between the two groups across time and within-subject observations of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged between 18 and 36
* Bilateral symptomatic flexible flatfoot, with symptoms including foot pain and lower limb fatigue
* Participants must show positive physical examination findings, including a positive result for the "too many toes" sign, the navicular drop test, and the foot toe raising test (Carr et al., 2016). A positive result for the "too many toes" sign occurs when more toes can be seen on the lateral side of each foot due to external rotation and abduction of the feet, and the positive result for the toe rising test is the reconstruction of the medial longitudinal arch secondary to the tightness of the plantar fascia (Carr et al., 2016). A positive result for the navicular drop test is an arch height more than or equal to 10 mm(Aenumulapalli et al., 2017)

Exclusion Criteria:

* An anatomical discrepancy in leg length
* Pathologic or neurologic disorders of the feet
* A history of traumatic foot injury or surgery within the last six months
* History of wearing foot orthoses within the past two years

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The EMED (force-area-pressure) | 6 weeks
  The feet plantar pressure was measured at baseline and at two-week intervals throughout the six-week intervention.

SECONDARY OUTCOMES:
Lower extremities functional scale, navicular drop test | 6 weeks
  The Lower extremities functional scale was used to evaluate restriction in participants' functional abilities, The score ranges from 0 to 80, and if it is higher indicating less functional restrictions. The navicular drop test was used to assess the medial longitudinal arch (MLA) height, A positive result for the navicular drop test is an arch height more than or equal to 10 mm. Both variables were measured at baseline and at the sixth week.

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastren, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Fattah, M.M., Hassanin, M.M., Felembane, F.A., Nassaane, M.T., 2006. Flat foot among Saudi Arabian army recruits: prevalence and risk factors. East. Mediterr. Health J. Rev. Sante Mediterr. Orient. Al-Majallah Al-Sihhiyah Li-Sharq Al-Mutawassit 12, 211-217. Abousayed, M.M., Tartaglione, J.P., Rosenbaum, A.J., Dipreta, J.A., 2016. Classifications in Brief: Johnson and Strom Classification of Adult-acquired Flatfoot Deformity. Clin. Orthop. 474, 588-593. Aenumulapalli, A., Kulkarni, M.M., Gandotra, A.R., 2017. Prevalence of Flexible Flat Foot in Adults: A Cross-sectional Study. J. Clin. Diagn. Res. JCDR 11, AC17-AC20. Allen, M.K., Glasoe, W.M., 2000. Metrecom Measurement of Navicular Drop in Subjects with Anterior Cruciate Ligament Injury. J. Athl. Train. 35, 403-406. Alnahdi, A.H., Alrashid, G.I., Alkhaldi, H.A., Aldali, A.Z., 2016. Cross-cultural adaptation, validity and reliability of the Arabic version of the Lower Extremity Functional Scale. Disabil. Rehabil. 38, 897-904. Aminian, G., Safaeepour, Z., Farhoodi, M., Pezeshk, A.F., Saeedi, H., Majddoleslam, B., 2013. The effect of prefabricated and proprioceptive foot orthoses on plantar pressure distribution in patients with flexible flatfoot during walking. Prosthet. Orthot. Int. 37, 227-232. Banwell, H.A., Mackintosh, S., Thewlis, D., 2014. Foot orthoses for adults with flexible pes planus: a systematic review. J. Foot Ankle Res. 7, 23. Buldt, A.K., Forghany, S., Landorf, K.B., Levinger, P., Murley, G.S., Menz, H.B., 2018. Foot posture is associated with plantar pressure during gait: A comparison of normal, planus and cavus feet. Gait Posture 62, 235-240. https://doi.org/10.1016/j.gaitpost.2018.03.005 Carr, J.B., Yang, S., Lather, L.A., 2016. Pediatric Pes Planus: A State-of-the-Art Review. Pediatrics 137, e20151230. Chen, Y.-C., Lou, S.-Z., Huang, C.-Y., Su, F.-C., 2010. Effects of foot orthoses on gait patterns of flat feet patients. Clin. Biomech. Bristol Avon 25, 265-270. Cheng, Y., Yang, H., Ni, L., Song, D., Zhang, H., 2015. Stress fracture of the distal fibula in flatfoot patients: case report. Int. J. Clin. Exp. Med. 8, 6303-6307. Chuter, V., Spink, M., Searle, A., Ho, A., 2014. The effectiveness of shoe insoles for the prevention and treatment of low back pain: a systematic review and meta-analysis of randomised controlled trials. BMC Musculoskelet. Disord. 15, 140. https://doi.org/10.1186/1471-2474-15-140 Daniels, T.R., Lau, J.T., Hearn, T.C., 1998. The effects of foot position and load on tibial nerve tension. Foot Ankle Int. 19, 73-78. https://doi.org/10.1177/107110079801900204 Dars, S., Uden, H., Kumar, S., Banwell, H.A., 2018. When, why and how foot orthoses (FOs) should be prescribed for children with flexible pes planus: a Delphi survey of podiatrists. PeerJ 6, e4667. https://doi.org/10.7717/peerj.4667 Giacomozzi, C., 2010. Appropriateness of plantar pressure measurement devices: A comparative technical assessment. Gait Posture 32, 141-144. https://doi.org/10.1016/j.gaitpost.2010.03.014 Hafer, J.F., Lenhoff, M.W., Song, J., Jordan, J.M., Hannan, M.T., Hillstrom, H.J., 2013. Reliability of plantar pressure platforms. Gait Posture 38, 544-548. https://doi.org/10.1016/j.gaitpost.2013.01.028 Hatfield, G.L., Cochrane, C.K., Takacs, J., Krowchuk, N.M., Chang, R., Hinman, R.S., Hunt, M.A., 2016. Knee and ankle biomechanics with lateral wedges with and without a custom arch support in those with medial knee osteoarthritis and flat feet. J. Orthop. Res. Off. Publ. Orthop. Res. Soc. 34, 1597-1605. https://doi.org/10.1002/jor.23174 Hegedus, E.J., Cook, C., Fiander, C., Wright, A., 2010. Measures of arch height and their relationship to pain and dysfunction in people with lower limb impairments. Physiother. Res. Int. 15, 160-166. https://doi.org/10.1002/pri.459 Hsieh, R.-L., Peng, H.-L., Lee, W.-C., 2018. Short-term effects of customized arch support insoles on symptomatic flexible flatfoot in children: A randomized controlled trial. Medicine (Baltimore) 97, e10655. https://doi.org/10.1097/MD.0000000000010655 Huang, Y.-C., Wang, L.-Y., Wang, H.-C., Chang, K.-L., Leong, C.-P., 2004. The relationship between the flexible flatfoot and plantar fasciitis: ultrasonographic evaluation. Chang Gung Med. J. 27, 443-448. Imhauser, C.W., Abidi, N.A., Frankel, D.Z., Gavin, K., Siegler, S., 2002. Biomechanical evaluation of the efficacy of external stabilizers in the conservative treatment of acquired flatfoot deformity. Foot Ankle Int. 23, 727-737.